CLINICAL TRIAL: NCT06557616
Title: Evaluation of the Safety and Efficacy of the CoolCryo System for Cardiac Cryoablation in the Treatment of Atrial Fibrillation in a Single-arm, Non-randomised, Open-label Clinical Trial
Brief Title: Safety and Efficacy of the CoolCryo System for Cardiac Cryoablation in the Treatment of Atrial Fibrillation
Acronym: CoolCryo
Status: Recruiting | Type: Observational
Sponsor: Medinice S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: BK_CIP-02
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation, Paroxysmal or Persistent; Mitral Valve Disease
Keywords: cryoablation; cardiac cryoablation; arrhythmia; atrial fibrillation; mitral valve; concomitant ablation
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The study involves endocardial cryoablation of the left and/or right atrium of the heart using the CoolCryo system as an adjunct to mitral valve surgery, with the aim of eliminating atrial fibrillation (AF), which is a common sequelae of mitral valve defects and is associated with an increased risk of ischaemic stroke, heart failure and death.

DETAILED DESCRIPTION:
An open-label, multi-centre, non-randomised study involving 16 patients, male and female, to evaluate the safety and efficacy of the CoolCryo system.

The procedure with the medical device will be performed on female and males aged ≥18 years, qualified for mitral heart valve surgery with a documented comorbidity of paroxysmal or persistent atrial fibrillation (AF) since at least 3 months prior to surgery excluding acute conditions.

The study involves endocardial cryoablation of the left and/or right atrium of the heart using the CoolCryo system as an adjunct to mitral valve surgery, with the aim of eliminating atrial fibrillation (AF), which is a common sequelae of mitral valve defects and is associated with an increased risk of ischaemic stroke, heart failure and death.

Data to assess the safety and efficacy of the CoolCryo system are collected at the time of the procedure and during the 6-month follow-up of the patient. In the clinical trial of the CoolCryo system, patient management at the Centre is conducted in accordance with the guidelines and standards of Polish and European medical societies, as well as taking into account the best practices developed at the Centre.

Due to the nature of the study population, 14 patients were taken as the minimum group size for which the CoolCryo device will be used. This size appears sufficient to analyse the safety and efficacy of the medical device used and was chosen for practical reasons and not on the basis of a formal sample size estimate. Given the 6-month follow-up period, the proportion of patients who will be lost to follow-up during the study was assumed to be 10 %. Therefore, 16 patients will be treated.

ELIGIBILITY:
Inclusion Criteria:

1. Written consent from the patient to participate in the study.
2. age ≥18 years.
3. patient qualified for mitral valve surgery (mitral valve plication or mitral valve replacement "with" or "without" left atrial appendage closure).
4. a documented diagnosis of co-occurrence of paroxysmal or persistent atrial fibrillation (AF) since at least 3 months prior to surgery with exclusion of acute conditions.

Exclusion Criteria:

1. Lack of written consent from the patient to participate in the study.
2. Failure to meet the inclusion criteria.
3. Contraindications to the cryoablation procedure.
4. Patient breastfeeding, pregnant or planning pregnancy within 6 months of study treatment.
5. co-morbidities and/or conditions that may cause atrial fibrillation (uncompensated hyperthyroidism or hypothyroidism, acute infection, pheochromocytoma, significant dyselectrolitemia).
6. significant calcification of the left atrium.
7. Condition after previous cardiac surgery.
8. significant left atrial enlargement (size greater than 10 cm on echocardiography in one of the projections performed). projection).
9. the patient is currently a participant in another clinical trial.
10. The patient is on active biological therapy.
11. emergency surgery.
12. Life expectancy <12 months.
13. Any circumstances that, in the opinion of the Investigator, may prevent the patient from participating in the study, limit the ability to perform the procedures outlined in the study protocol or place an unreasonable risk on the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sixteen patients, male and female, aged ≥18 years, qualified for mitral heart valve surgery with documented (in at least one ECG recording) co-occurrence of paroxysmal or persistent atrial fibrillation (AF) will undergo the procedure with the medical device.
  There is also a prediction of 10 per cent of patients (screen failure) who do not meet the inclusion and/or exclusion criteria after signing informed consent.
  Additionally, there may be perioperative situations where the cryoablation procedure is not performed due to potential acute aortic dissection or undiagnosed conditions necessitating a change in surgical tactics (e.g. pericarditis). It is estimated that the above situation may affect 1-2 study participants who will be given drop-out status.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with no documented recurrence of atrial fibrillation on continuous 48h Holter ECG recording during 6-month follow-up. | 12 weeks (+/- 7 days) and 25 weeks (+/- 7 days) after the procedure
  To verify whether atrial fibrillation is present in the recordings obtained during 48h Holter. ECG monitorin
Incidence of adverse events and serious adverse events related to the use of the | 6 day (+/- 1 day), 12 weeks (+/- 7 days) and 25 weeks (+/- 7 days) after the procedure
  Recording of adverse events/serious life-threatening events.

SECONDARY OUTCOMES:
The occurrence of serious adverse events during surgery (intraoperatively) or after the procedure until the patient is discharged from the unit (postoperatively). | During the procedure, 6 day (+/- 1 day) after the procedure
  Recording of all adverse events/serious life-threatening events.
Incidence of all adverse events and serious adverse events at 6-month follow-up after surgery. | 6 day (+/- 1 day), 12 weeks (+/- 7 days) and 25 weeks (+/- 7 days) after the procedure
  Recording of all adverse events/serious life-threatening events.
The proportion of patients who had a return to sinus rhythm at 3 and 6 months postoperatively. | 12 weeks (+/- 7 days) and 25 weeks (+/- 7 days) after the procedure
  To verify whether sinus rhythm is present in the recordings obtained during 48h Holter ECG monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Hrapkowicz, MD PhD, Principal Investigator — Silesian Centre for Heart Diseases
Locations (2):
- Poland (2):
  - Antoni Jurasz University Hospital No. 1, Bydgoszcz
  - Silesian Centre for Heart Diseases, Zabrze